CLINICAL TRIAL: NCT03670004
Title: Sensory-Motor Mechanisms Underlying Fall Risk in Transtibial Amputees
Brief Title: Falls in Older Persons With Limb Loss
Acronym: FOPLL
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C1322-W; IK2RX001322 (NIH)
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-04

CONDITIONS: Amputation; Elderly
Keywords: Artificial Limbs; Amputation; Accidental Falls; Stability; Balance; Gait; Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Unilateral Below Knee Amputation: Individuals who walk with a below knee prosthesis
- Non-Impaired: Able-bodied controls

SUMMARY:
Lower limb prosthesis users are known to be at a substantially increased fall risk compared to able-bodied individuals. The interaction between increased fall risk, reduced balance confidence and high prevalence of a fear of falling often leads to restricted mobility and loss of independence. Critically, the cause of these falls and the role that inherent balance plays in fall risk is poorly understood. This study proposes to identify key differences in balance and mobility between older below-knee prosthesis users and able-bodied individuals. By further understanding the differences between these groups and relationships between fall risk and various outcome measures, intervention techniques can be developed to improve functional balance. An improvement in upright balance will reduce the occurrence of falls and fall related injuries in this veteran population, as well as increase their participation in daily activities and improve their quality of life.

DETAILED DESCRIPTION:
Previous studies have shown that persons with transtibial amputations (TTA) are at a substantially increased risk of falling as compared to able-bodied age-matched controls and have reduced confidence in their balance, both contributing to their restricted mobility and daily activity. This risk increases with progressing age, as aging affects musculoskeletal and somatosensory systems that are vital to controlling upright balance (i.e., maintaining the body center-of-mass (BCoM) within the limits of the base-of-support) and are already compromised in persons with TTA. An important consequence of elevated fall incidence is an increased risk of fall-related injuries that may lead to lost participation and independence. The effects of reduced sensory-motor function on upright balance in older adults has been extensively studied and led to development of effective assessment tools and intervention strategies to minimize fall risk. However, the dearth of similar studies and relatively poor understanding of the effects of additional complications from TTA on upright balance have significantly hampered progress towards addressing this important concern for Veterans with TTA. Consequently, this limits knowledge of predictive factors of falls among these prosthesis users and for informing therapeutic interventions that enhance functional balance. Therefore, the primary objective of this research is to develop an improved understanding of the sensory-motor mechanisms underlying upright balance and fall risk in older Veterans with TTA. The proposed study will compare differences between two age- and gender-matched groups: 1) older unilateral prosthesis users and 2) able-bodied controls.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the recruitment of subjects with below knee amputation include:

* Transtibial amputation
* Daily use of their clinically-prescribed prosthesis for ambulation without an assistive device
* Classified as Medicare Functional Classification Level K2- defined as a patient who "has the ability or potential for ambulation with the ability to traverse low-level environmental barriers such as curbs, stairs, or uneven surfaces - a typical community ambulator"
* Experience walking with a prosthesis for at least one year
* Residuum and amputated side in good condition (e.g., no adherent scars, lesions, ulcers, infections)
* Normal or corrected vision
* Able to walk a 10 m distance and stand quietly for 40 seconds without undue fatigue or health risk

Inclusion criteria for the recruitment of able-bodied controls include:

* Normal or corrected vision
* Able to walk a 10 m distance and stand quietly for 40 seconds without undue fatigue or health risk
* Suffered one or no falls in the previous 12 months

Exclusion Criteria:

Exclusion criteria for all recruited subjects (i.e., limb loss and control) include:

* Musculoskeletal (apart from amputation in the case of amputee subjects) and/or vestibular pathologies that would affect balance and/or stability
* Currently on medication that might affect proprioception and/or balance (e.g., drugs that are ototoxic, such as certain Aminoglycosides and pain killers)
* Cognitive deficits that preclude understanding of the instructions required to conduct the test

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older ambulatory individuals with or without unilateral below-knee amputation
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Major, PhD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unilateral Below Knee Amputation | Non-Impaired
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unilateral Below Knee Amputation | Non-Impaired | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (3.8) | 71.7 (4.2) | 71.4 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 10 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Foot's Height During the Swing Phase of Walking (i.e., Foot Clearance) Measured in Centimeter
Description: Foot clearance of self-selected normal and fast speed walking, calculated as the distance (cm) between the toe and ground as measured with an optical motion capture system.
Time Frame: 1 month
Population: Foot clearance was measured for each limb at each walking speed
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Limbs
Arm/Group | Unilateral Below Knee Amputation | Non-Impaired
Number analyzed (Participants) | 13 | 10
Number analyzed (Limbs) | 26 | 20
cm
  Non-dominant/Impaired, normal speed | 6.1 (1.5) | 5.5 (1.2)
  Dominant/Sound, normal speed | 6.1 (1.3) | 5.7 (1.3)
  Non-dominant/Impaired, fast speed | 5.1 (1.2) | 4.1 (0.8)
  Dominant/Sound, fast speed | 4.7 (0.7) | 4.2 (0.9)

2. Primary Outcome: Center of Pressure Sway Area During Eyes Open or Closed as Measured Through a Force Plate During Standing and Calculated as Centimeters Squared
Description: Center of pressure sway area during eyes open or closed, calculated as the area (cm*cm) covered by the center of pressure position during standing as measured with a force plate.
Time Frame: 1 month
Population: Sway area was measured for each limb for each vision condition of eyes open or closed
Measure: Mean (Standard Deviation); unit: cm*cm
Units Other Than Participants: limbs
Arm/Group | Unilateral Below Knee Amputation | Non-Impaired
Number analyzed (Participants) | 13 | 10
Number analyzed (limbs) | 26 | 20
cm*cm
  Dominant/Sound, eyes open | 1.26 (1.12) | 0.99 (1.39)
  Non-dominant/Impaired, eyes open | 0.66 (0.48) | 0.71 (0.67)
  Dominant/Sound, eyes closed | 1.22 (0.94) | 0.79 (0.80)
  Non-dominant/Impaired, eyes closed | 0.64 (0.43) | 0.76 (0.81)

3. Primary Outcome: Gait Muscle Activation Effort as Measured by Sensors and Integrating Measured Voltage With Respect to Time as to be Calculated as Millivolts Times Seconds
Description: Integrated Electromyography patterns of leg muscles during self-selected normal and fast speed walking as a proxy measure of muscle effort, calculated from integrating the muscle activity measured by sensors as voltage over time (mv*sec)
Time Frame: 1 month
Population: Integrated EMG was measured for each muscle group of interest at each walking speed
Measure: Mean (Standard Deviation); unit: mv*sec
Units Other Than Participants: Muscle group
Arm/Group | Unilateral Below Knee Amputation | Non-Impaired
Number analyzed (Participants) | 13 | 10
Number analyzed (Muscle group) | 26 | 20
mv*sec
  Dominant/Sound Tibilias Anterior, normal speed | 0.278 (0.069) | 0.306 (0.067)
  Dominant/Sound Tibilias Anterior, fast speed | 0.372 (0.096) | 0.348 (0.098)
  Dominant/Sound Gastroc, normal speed | 0.360 (0.041) | 0.256 (0.079)
  Dominant/Sound Gastroc, fast speed | 0.307 (0.063) | 0.318 (0.123)

4. Secondary Outcome: Falls
Description: Number of falls during 12 months prospectively
Time Frame: 1 year
Population: Total number of falls 12 months prospectively
Measure: Number; unit: Falls
Arm/Group | Unilateral Below Knee Amputation | Non-Impaired
Number analyzed (Participants) | 13 | 10
Falls | 18 | 10

ADVERSE EVENTS:
Time Frame: 12 months prospectively
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Unilateral Below Knee Amputation | Non-Impaired
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unilateral Below Knee Amputation (N=13) | Non-Impaired (N=10)
Head Injury (General disorders) | 1 (1) | 0 (0) — Head injury experienced from a fall during 12-month prospective fall data collection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT03670004/Prot_SAP_000.pdf